CLINICAL TRIAL: NCT06801093
Title: Evaluating the Impact of a Digital Psychosocial Tool (Wysa) on Life Skills and Overall Well-being With English-Speaking College Students in Gandhinagar, India: A Mixed Methods Feasibility Study
Brief Title: Evaluating the Impact of a Digital Psychosocial Tool (Wysa) on Life Skills and Well-being of College Students in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: Wysa (Industry)
Responsible Party: Principal Investigator, Sarah Jasim, Research Fellow, London School of Economics and Political Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 390706
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-01

CONDITIONS: Wellbeing; Resilience; Self Efficacy; Life Skills; Problem Solving
Keywords: digital psychosocial tool; wellbeing; life skills; college student; digital intervention; feasibility study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wysa app (Experimental): Participants will receive the digital psychosocial tool (Wysa) for a period of 2 months. Wysa is a digital app that includes an AI-based conversational conversational agent, a repository of self-help tools, and SOS resources.
  Interventions: Behavioral: Digital psychosocial tool

INTERVENTIONS:
Behavioral: Digital psychosocial tool — Wysa is a digital psychosocial tool that provides AI conversational chatbot support. The conversational agent acts as a companion, and understands, empathizes, and guides users through exercises grounded in cognitive behavioral therapy (CBT), mindfulness, and motivational intervention. Participants can progressively work through learning different skills and practice them in their daily life. The app also provides a repository of tools to manage problems and SOS resources for high distress.

SUMMARY:
The goal of this study is to learn the feasibility of a digital psychosocial tool (Wysa) in improving life skills and overall wellbeing of English-speaking college students in IIT-Gandhinagar, a university in India. This will be conducted using pre-post assessments examining resilience, self-efficacy, problem solving, and wellbeing as well as examining app usage during the intervention period. The main questions it aims to answer are:

1. The feasibility and acceptability of Wysa amongst college students enrolled at the university
2. The effectiveness of Wysa in improving the life skills and well-being of college students enrolled at the university

DETAILED DESCRIPTION:
This study will employ a mixed methods pre-post design to examine whether a digital psychosocial tool can help college students in India learn ways to manage their problems and improve their wellbeing. Students enrolled at the Indian Institute of Technology, Gandhinagar (IIT-Gn) and are interested in learning skills to manage stressors are invited to participate in the study. The intervention being studied is the Wysa app which includes an AI-based chatbot, a library of toolpacks , and SOS resources. Participants will complete baseline research procedures (T0) and be able to download the app. Participants can use the Wysa app for a period of 2 months. At the end of 2 months, participants will be invited to complete their endline assessments (T1). Another follow-up assessment (T2) will be carried out 1 month after the intervention period completion. A sub-sample of participants will be invited to participate in qualitative interviews to provide feedback about their experiences using the Wysa app and to understand the barriers and facilitators to acceptability and effectiveness of the app.

ELIGIBILITY:
Inclusion Criteria:

* Are between 18-25 years of age
* Are a student of Idian Institute of Technology, Gandhinagar (IIT Gandhinagar)
* Are able to read and understand English
* Have access to an internet enabled smartphone

Exclusion Criteria:

* Have previously used Wysa app (the intervention)
* Presence of self-harm/suicidal risk

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment rate | Measured during the recruitment period (1 month, or if recruitment is extended at the end of 2 months)
  Proportion of participants who completed consent procedures
Feasibility - Retention rate | Measured after the 2 month intervention during follow-up assessments
  Proportion of recruited participants who completed endline assessments and follow-up assessments i.e. those who remained enrolled for the study duration.
Feasibility - App onboarding rate | Measured during the 2 month intervention period
  Proportion of participants who downloaded the app after allocation to the intervention
Acceptability - Wysa app engagement | Measured during the 2-month intervention period
  Proportion of recruited participants who interacted with Wysa at least once after onboarding to the app. Information will also collected on average numbers of days the app was used. Analysis of usage of different app features and tools will also be conducted.
App satisfation | This is collected thrice during the 2-month intervention period
  Feedback is collected through questions which ask participants to provide a quantitative rating of the app features' usability and satisfaction. Participants can provide ratings on a 5 point likert scale with higher ratings denoting higher satisfaction. 1 qualitative question invites participant to use free text format to provide any additional feedback.
App Acceptability and experiences of usage | Conducted after the intervention period (2 months)
  Semi-structured interviews with a sub-sample of participants will provide insights into the lived experience of using the intervention; and barriers and facilitators to usage.

SECONDARY OUTCOMES:
Changes in wellbeing as measured on the WHO Wellbeing Index | 3 months: at Month 0 (pre-intervention), Month 2 (post-intervention period), Month 3 (1-month after intervention period)
  The WHO Wellbeing Index is a 5-item questionnaire assessing an individual's wellbeing. Participants can respond to how frequently they have felt the item asked on a 6-point likert scale. Scores range from 0-25
Changes in problem solving as measured on the Problem Solving Inventory | 3 months: at Month 0 (pre-intervention), Month 2 (post-intervention period), Month 3 (1-month after intervention period)
  The Problem Solving Inventory (PSI) is a 35-item scale. Participants can provide a rating of their problem solving skills on a 6-point likert scale from strongly agree to strongly disagree. The scale provides a score range from 35-210.
Changes in self-efficacy as measured on the general self-efficacy scale | 3 months: at Month 0 (pre-intervention), Month 2 (post-intervention period), Month 3 (1-month after intervention period)
  The General Self-Efficacy Scale is a 10-item scale. Participants can rate their self-efficacy on a 4-point likert scale ranging from 'not at all true' to 'exactly true'. The scale provides a score range between 10-40.
Changes in resilience, as measured on the Brief Resilience Scale | 3 months: at Month 0 (pre-intervention), Month 2 (post-intervention period), Month 3 (1-month after intervention period)
  The Brief Resilience Scale (BRS) includes 6 items and assesses an individual's ability to bounce back from stressors. Scores on each item range from 1-5 for with all six items giving a range from 6-30.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jasim, Ph.D, Principal Investigator — London School of Economics and Political Science
Locations (1):
- Indian Institute of Technology, Gandhinagar (IIT-Gandhinagar), Palaj, Gujarat, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any external party as it does not comply with the terms of consent.